CLINICAL TRIAL: NCT01910233
Title: Prospective Registry for Quality Assurance of Medical Care of Patients With Acute Dyspnea in the Emergency Department
Brief Title: Registry of Patients With Acute Dyspnea in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Christ, Prof. Dr. med. Michael Christ, Klinikum Nürnberg
Other Study IDs: OOB01
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Dyspnea; Heart Failure; COPD
Keywords: dyspnea; registry; baseline characteristics; mortality; risk assessment; emergency department
MeSH Terms: conditions — Dyspnea; Heart Failure; Pulmonary Disease, Chronic Obstructive; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adult patients with acute dyspnea in ED

SUMMARY:
This is a prospective registry of patients presenting with acute dyspnea to the emergency department of the city hospital in Nuremberg. There is evidence that acute dyspnea is associated with a mortality rate of 10%, however acute dyspnea is not perceived as a life-threatening condition, both in public and in health care providers. Our aim is to describe the patient collective concerning their demographics, baseline characteristics, type of referral and disposition, medical care processes and prognosis. Secondly, we want to evaluate if the subjective risk assessment of emergency department personnel matches with objective risk stratification tools and the actual outcome of the studied patients.

DETAILED DESCRIPTION:
This is a prospective registry of patients presenting with acute dyspnea to the emergency department of the city hospital in Nuremberg during May 23th 2013 and October 31th 2013. To be included into the registry the patient has to express acute dyspnea. Minor patients are not included. The admission documents of the studied patients are accompanied by a questionnaire that has to be completed by the triage nurse and the attending physician. The questionnaire includes items like professional experience and subjective assessment of patient's prognosis. In addition the attending physician has to state if the evaluation of medical history was difficult, if previous medication is known and how likely the presence of heart failure as underlying condition is. Data of the questionnaire, the patient record and the follow up contacts are entered in a SPSS database. Finally, we measure the OPTIMIZE-HF score (Abraham et al. 2008) and the PRIDE mortality score (Baggish et al. 2007) in a retrospective manner in order to compare the subjective assessments with objective criteria.

ELIGIBILITY:
Inclusion Criteria:

* expression of acute dyspnea in the emergency department

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department of the city hospital Nuremberg
Sampling Method: Probability Sample
Enrollment: 947 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 6 months

SECONDARY OUTCOMES:
demographics and baseline characteristics | 1 month
  baseline characteristics as for example vital signs, medication, underlying disease condition (adjusted final diagnosis), medical history, concomitant diseases
medical care processes | 1 day
  type of referral, disposition patterns, diagnostic and therapeutical measures
subjective and objective risk assessment | 1 month
  data from the questionnaire completed by triage nurse and attending physician, OPTIMIZE-HF and PRIDE mortality score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Christ, Prof., Principal Investigator — Klinikum Nürnberg
Locations (1):
- Department of Emergency and Critical Care Medicine, City Hospital Nuremberg, Nuremberg, Bavaria, Germany